CLINICAL TRIAL: NCT06106295
Title: Metyrapone Intervention in Patients With Mild Autonomous Cortisol Secretion (MACS)
Brief Title: Metyrapone for Mild Autonomous Cortisol Secretion (MACS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Irina Bancos, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-008085
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Autonomous Cortisol Secretion; Mild Autonomous Cortisol Secretion (MACS)
Keywords: Hypercortisolism; Cortisol excess; Cushing syndrome; Adrenal adenoma; Adrenal hyperplasia
MeSH Terms: conditions — Cushing Syndrome; ACTH Syndrome, Ectopic; Adrenal Hyperplasia, Congenital | interventions — Metyrapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mild Autonomous Cortisol Secretion (MACS) Open Label Phase and Optional Extension Phase (Experimental): Subjects diagnosed with Mild Autonomous Cortisol Secretion (MACS) will receive metyrapone for a 6 month treatment period (Open Label Phase) with the option to continue for an additional 30 months of metyrapone therapy. If a patient chooses to participate in the Optional Extension Phase they will continue to receive metyrapone therapy until Month 36. This is an additional 30 months of therapy after completion of the Open Label Phase.
  Interventions: Drug: Metyrapone

INTERVENTIONS:
Drug: Metyrapone — 250 to 1000 milligram (mg) orally in one or two doses in the evening (administered 4 and 2 hours prior to bed)

SUMMARY:
The purpose of this study is to find out whether the study drug, metyrapone, is safe and effective in treating participants with Mild Autonomous Cortisol Secretion (MACS).

DETAILED DESCRIPTION:
This study will look at how well metyrapone controls blood pressure, blood glucose, blood lipids and weight.

Metyrapone is approved in the United States of America (USA) by the Federal Drug Administration (FDA) for use in the diagnosis of adrenal insufficiency. It is not approved in the USA for the treatment of MACS. It is approved in Europe for the treatment of ACTH dependent Cushing's Syndrome.

Metyrapone is currently being tested to evaluate the safety (side effects/risks) and efficacy (benefits), so its use for the treatment of MACS is experimental in the USA. Its effectiveness is unproven in the USA and metyrapone is considered an investigational study drug in the USA. The Mayo Clinic IRB has given approval for this drug to be used in this setting.

Patients diagnosed with MACS have abnormal cortisol levels above the normal range. Cortisol acts by binding with the cortisol receptors in many tissues of the body. Metyrapone works by reducing cortisol production, thereby decreasing the effects of too much cortisol. Metyrapone doesn't affect levels of other hormones in your body.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Diagnosed with MACS: at least 2 abnormal post-dexamethasone cortisol results (1 mg post-dexamethasone cortisol > 1.8 mcg/d; or 8 mg post-dexamethasone cortisol > 1 mcg/dL) and historical dexamethasone suppression test results can be used if performed within 24 months prior to enrollment.
* Adrenal imaging phenotype consistent with benign disease (adrenal adenoma/s, macronodular or micronodular adrenal hyperplasia).
* At least one of the following comorbidities: obesity (BMI > 30 kg/m^2); dysglycemia; dyslipidemia; hypertension; osteopenia; osteoporosis; fragility fractures.
* Ability to take oral medication and be willing to adhere to the study intervention regimen.
* For females of reproductive potential: use of highly effective contraception initiated prior to baseline visit and for 1 month after completing metyrapone study.
* For persons of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of <5% per year during the treatment period and for 6 months after the last dose of study treatment.
* Stable timing for bedtime for at least one week prior to on-site study visits

Exclusion Criteria:

* Planned alternative therapy for MACS within 6 months after joining the study.
* Current use of oral exogenous glucocorticoid therapy.
* Current use of opioid therapy > 20 MME/day.
* Planned use of oral exogenous glucocorticoid therapy.
* Planned use of opioid therapy > 20 MME/day.
* Use of injectable glucocorticoid within the last 6 weeks.
* Investigator's judgement based on history/physical examination that a comorbidity or concomitant medication may impact the hypothalamic-pituitary-adrenal axis or steroid metabolome.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnancy or lactation.
* Known allergic reactions to metyrapone.
* Suspected false positive post-dexamethasone cortisol results due to increased metabolism, poor absorption, or noncompliance with dexamethasone.
* Treatment with another investigational drug or other intervention within lower than specific therapy washout period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 50 months
  Number of participants to experience adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Irina Bancos, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials